CLINICAL TRIAL: NCT04018560
Title: Intensive Referral to Al-Anon: Benefits to Concerned Others and Their Drinkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Veterans Institute for Research (Other)
Responsible Party: Principal Investigator, Christine Timko, Principal Investigator, Palo Alto Veterans Institute for Research
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: TIM0026
Record Dates: First submitted 2019-07-08; First posted 2019-07-12 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Al-Anon Intensive Referral (AIR)
- Usual care (No Intervention)

INTERVENTIONS:
Behavioral: Al-Anon Intensive Referral (AIR) — AIR is intended to facilitate Al-Anon participation.
  Arms: Intervention

SUMMARY:
This study is examining the effectiveness of Al-Anon Intensive Referral (AIR) with Concerned Others (COs) of individuals in treatment for alcohol use disorders ("drinkers"). AIR's goal is to facilitate Al-Anon participation and positive outcomes among COs.

DETAILED DESCRIPTION:
In a randomized controlled trial, this 4-year project is evaluating AIR's effectiveness for COs. COs and their drinkers are assessed at baseline and 3-month, 6-month, and 1-year follow-ups. Hypotheses are that, compared to usual care, AIR will increase Al-Anon participation and improve CO outcomes. We will examine hypotheses using generalized mixed-effects regression models (GLMM). This project is built on the foundation that it is essential to help COs because of their own suffering.

ELIGIBILITY:
Inclusion Criteria:

1. the drinker is an adult (≥19 years old) entering a treatment episode for the primary substance of alcohol;
2. the drinker signs a release for researchers to contact a CO (also an adult) he or she identifies as a family member or close friend who has had contact with the drinker on at least 12 (40%) of the past 30 days; and
3. the drinker and CO can communicate in English. -

Exclusion Criteria:

1. the drinker is <19 years old, not entering a treatment episode for alcohol use disorder;
2. the drinker does not sign a release for researchers to contact a CO;
3. the drinker and CO cannot communicate in English. -

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Mental Health | The outcome measure will be assessed up to 1 year follow-up.
  Items are rated on a 5-point scale (0=never, 4=very often). Mental Health is the mean of 10 items (e.g., How often have you experienced feeling hopeful); negative symptoms (e.g., anxious) are reverse scored.

CONTACTS AND LOCATIONS:
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

REFERENCES:
- [Derived] Timko C, Cucciare MA, Lor MC, Stein M, Vest N. Patient-Concerned Other Dyads' 12-Step Involvement and Patients' Substance Use: A Latent Class Growth Model Analysis. J Stud Alcohol Drugs. 2023 Sep;84(5):762-771. doi: 10.15288/jsad.22-00378. Epub 2023 May 18. PMID 37219032
- [Derived] Timko C, Grant KM, Han X, Young LB, Cucciare MA. Al-Anon Intensive Referral to facilitate concerned others' participation in Al-Anon Family Groups: a randomized controlled trial. Addiction. 2022 Mar;117(3):590-599. doi: 10.1111/add.15670. Epub 2021 Oct 3. PMID 34427006